CLINICAL TRIAL: NCT05247931
Title: Why Does Aspirin Fail in Secondary Cerebrovascular Prevention? A Multicenter Prospective Case - Control Study
Acronym: ASTRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.01.2018
Record Dates: First submitted 2022-01-20; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE: patients experiencing a recurrent stroke while on ASA therapy
  Interventions: Diagnostic Test: TXB2 assay of serum , and 11-dehydro-TXB2 assay of urine
- CONTROL: ASA-naïve patients experiencing a first atherothrombotic stroke
  Interventions: Diagnostic Test: TXB2 assay of serum , and 11-dehydro-TXB2 assay of urine

INTERVENTIONS:
Diagnostic Test: TXB2 assay of serum , and 11-dehydro-TXB2 assay of urine — Blood samples are analyzed for the assay of serum TXB2, and urine samples for the assay of 11-dehydro-TXB2

SUMMARY:
Multicenter prospective observational case-control study aimed at characterizing the possible determinants of treatment failure in patients with cerebrovascular disease on secondary prevention with ASA, who are hospitalized in Internal Medicine departments for a recurrent atherothrombotic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Swallow-test positive
3. Patients hospitalized for a first event of athero-thrombotic stroke (CONTROL group)
4. Patients hospitalized for a recurrence of athero-thrombotic stroke on ASA therapy (CASE group)
5. Informed Consent

Exclusion Criteria:

1. Transient ischemic attack (TIA)
2. Chronic treatment with non-steroidal anti-inflammatory drugs (if occasional, not within 4 days prior to hospitalization)
3. Current treatment with oral or parental anticoagulants at prophylactic or therapeutic doses
4. Current treatment with other antiplatelet agents
5. Thrombolysis and thrombectomy
6. Cardio-embolic stroke CENTRO STUDI FONDAZIONE FADOI Page 10 Studio FADOI.01.2018 Versione n. 2 del 26/09/2019
7. Carotid stenosis >70%, with indication for revascularization
8. Current treatment with ASA (only for patients in the CONTROL group)
9. Acute hepatitis, chronic active hepatitis, liver cirrhosis - or alanine aminotransferase level 3 times or more and/or bilirubin level 2 times or more higher than the upper limit of the normal range
10. Thrombocytopenia (<150000 platelets/μl)
11. Renal failure (eGFR <30 ml/min)
12. Active cancer or disease in complete remission <1 year, except squamous cell carcinoma and basal-cell carcinoma of the skin at initial stage
13. Severe chronic obstructive pulmonary disease (COPD) (oxygen therapy)
14. Uncontrolled hypertension (systolic BP >180 mmHg or diastolic BP >100 mmHg despite antihypertensive treatment)
15. Chronic inflammatory bowel disease
16. Chronic treatment with corticosteroid drugs (for example Prednisone >5 mg/die or equivalent)
17. Pregnancy (in case of child-bearing potential inclusion will be possible in case of negative pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with athero-thrombotic stroke, to be divided into CASE group (50 patients experiencing a recurrent stroke while on ASA therapy) and CONTROL group (50 ASA-naïve patients experiencing a first atherothrombotic stroke), with ratio 1:1.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of recovery of platelet COX-1 activity, measured between 12 and 24 hours after low-dose (100 mg) ASA administration by means of three determinations of serum TXB2 levels, at day 8±1, comparing CASE group vs. CONTROL Group. | day 8±1
  To evaluate the rate of recovery of platelet COX-1 activity, measured between 12 and 24 hours after low-dose (100 mg) ASA administration by means of three determinations of serum TXB2 levels, at day 8±1, comparing CASE group vs. CONTROL Group.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA FONTANELLA, Study Director — FONDAZIONE FADOI
Locations (16):
- Italy (16):
  - Ospedale di Assisi, Assisi
  - Ospedale Maggiore di Bologna, Bologna
  - Ospedale "S. Cuore di Gesù" Gallipoli, Gallipoli
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Di Mantova, Mantova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - P.O. Ostuni-Fasano - ASL BR, Ostuni
  - IRCCS Mondino, Pavia
  - Azienda Ospedaliera Santa Maria della Misericordia, Perugia
  - Ospedale di Pordenone, Pordenone
  - Policlinico Gemelli, Roma
  - Ospedale Umberto I - ASP Siracusa, Syracuse
  - Ospedale Molinette, Torino
  - Ospedale Ca' Foncello di Treviso, Treviso
  - Ospedale di Circolo -ASST Settelaghi, Varese
  - Ospedale Dei Colli, Viterbo

IPD SHARING:
Plan to Share IPD: Undecided